CLINICAL TRIAL: NCT05251064
Title: Randomized Controlled Trial of Wound Closure Techniques in Orthopaedic Surgery
Brief Title: Orthopaedic Surgical Wound Closure Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21411
Record Dates: First submitted 2022-01-21; First posted 2022-02-22 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Incision, Surgical
MeSH Terms: conditions — Surgical Wound | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Suture (Active Comparator): Standard suture wound closure
  Interventions: Device: Suture
- Adhesive wound closure device (Active Comparator): Clozex wound closure device
  Interventions: Device: Clozex
- Adhesive wound closure device with zip ties (Active Comparator): Zipline wound closure device
  Interventions: Device: Zipline

INTERVENTIONS:
Device: Suture — Standard suture wound closure device.
  Arms: Suture
Device: Clozex — Interlaced adhesive wound closure device.
  Arms: Adhesive wound closure device
Device: Zipline — Adhesive wound closure device using zip-tie like strips.
  Arms: Adhesive wound closure device with zip ties

SUMMARY:
This study is trying to find out if there is one method of surgical incision closure is better than another. The three different wound closure methods in this study are currently used in standard of care. The three methods being compared are standard stitches and the wound closure devices, Clozex, and Zipline. All of these methods are approved by the FDA.

DETAILED DESCRIPTION:
There are many surgical wound closure methods commonly used in practice today. These usually involve a combination of braided and monofilament sutures in the subcutaneous fascia and fat as well as the subcuticular layers of the skin. The methods chosen by surgeons vary widely even amongst partners at the same institution for many reasons, including training background and conflicting reports in the literature. In some cases, these closure techniques can be time consuming and associated with increased rates of poor cosmetic outcomes or complications. There have been new wound closure products to reach the market that have been designed (Zipline - Campbell, CA and Clozex - Wellesley, MA), claiming to increase the speed of closure and decrease the rate of complications. These products both utilize an adhesive backed film to adhere to the skin along with a proprietary method to enhance skin apposition to reduce tension during the healing process. There has been no randomized controlled trial to determine superiority of the above listed surgical closure methods compared to traditional methods.

Our study aims to compare a "traditional" wound closure using both braided and monofilament sutures to the newer wound closure systems. By determining which method provides superior results, we will improve patient outcomes and satisfaction. The study also aims to assess health care value by exploring the costs associated with each closure technique. In addition to material expenses associated with the traditional sutures, we seek to explore if there is a significant difference in the time required to perform each wound closure method. Every minute of anesthesia and operating room utilization is associated with costs borne by the patient and the health care system. By finding which closure method is the fastest and associated with the best outcome we can improve healthcare value.

These methods will be tested in a randomized controlled trial and will be analyzed with multivariate statistical analysis to examine statistical significance. Subjects will be randomized in a 1:1:1 fashion to sutures, Closex, or Zipline. Surgeons will complete a satisfaction questionnaire about the randomized method used for closure. Surgical subjects will complete a satisfaction questionnaire at two follow up visits that align with standard of care visits and will have the incision measured and examined. Our primary objective outcome measure will be an assessment of surgical scar dimensions. Our hypothesis is that the 3 study groups will have similar objective scar measurements but that the savings in time associated with the new wound closure methods will be significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Patient scheduled to undergo elective orthopaedic surgical procedure with a minimum anticipated incision length of 3 cm.
* Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

* Revision Surgery
* Compromised wound healing (autoimmune disorder, chronic steroids, connective tissue disorder)
* Pregnant women, fetuses, neonates, children, prisoners, cognitively impaired, educational or economically disadvantage, non-English speaking subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Miller, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be share. Group means will be shared.

REFERENCES:
- [Derived] Burke JF, MacLean IS, Smith JM, Hart JM, Miller MD. A Prospective, Randomized, Controlled Comparison of Adhesive Wound Closure Devices in an Orthopaedic Patient. J Am Acad Orthop Surg Glob Res Rev. 2022 Sep 23;6(9):e22.00179. doi: 10.5435/JAAOSGlobal-D-22-00179. eCollection 2022 Sep 1. PMID 36155955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Started | 19 | 19 | 18
Completed | 10 | 11 | 11
Not Completed | 9 | 8 | 7

BASELINE CHARACTERISTICS:
Population: This is the number of subjects included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties | Total
Number analyzed (Participants) | 10 | 11 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 11 | 31
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (18.5) | 40.9 (10.6) | 34.6 (16.7) | 38.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 19
  Male | 4 | 5 | 4 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: Stony Brook Scar Evaluation Scale
Description: Scores range from 0-5. Higher scores indicate better scar healing. Lower scores indicate worse scar healing
Time Frame: 2-Weeks post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
score on a scale | 2.8 (0.92) | 4.09 (0.70) | 3.45 (1.21)

2. Primary Outcome: Stony Brook Scar Evaluation Scale
Description: Scores range from 0-5. Higher scores indicate better scar healing. Lower scores indicate worse scar healing
Time Frame: 3-Months post operative
Population: All subjects who completed 3-Month follow-up and were randomized to their respective wound closure device.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
score on a scale | 2.85 (1.20) | 3.82 (0.60) | 3.0 (0.89)

3. Secondary Outcome: Time to Close
Description: The amount of time in seconds that it took to perform closure of the incision.
Time Frame: During the procedure, from beginning of wound closure to the completion of wound closure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
seconds | 266.31 (193.59) | 91.09 (39.53) | 123.27 (124.23)

4. Secondary Outcome: Length of Incision
Description: This is the measure in centimeters of the incision.
Time Frame: During the procedure, obtained after incision was closed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
centimeters | 9.78 (4.87) | 8.23 (4.09) | 8.1 (2.78)

5. Secondary Outcome: Patient Satisfaction
Description: Scores range from 0-10. Higher scores indicate better satisfaction. Lower scores indicate lower patient satisfaction.
Time Frame: 2 weeks post operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
units on a scale | 8.33 (1.66) | 8.82 (1.33) | 8.64 (1.8)

6. Secondary Outcome: Patient Satisfaction
Description: Scores range from 0-10. Higher scores indicate better satisfaction. Lower scores indicate lower patient satisfaction.
Time Frame: 3 months post operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
units on a scale | 8.11 (1.95) | 8.727 (1.73) | 8.82 (1.47)

7. Secondary Outcome: Surgeon Satisfaction
Description: Scores range from 0-10. Higher scores indicate better satisfaction. Lower scores indicate lower satisfaction.
Time Frame: Once (at application)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
Number analyzed (Participants) | 10 | 11 | 11
units on a scale | 7.11 (3.62) | 8.18 (2.09) | 8.0 (1.55)

ADVERSE EVENTS:
Time Frame: 3 months.
Arm/Group | Suture | Adhesive Wound Closure Device | Adhesive Wound Closure Device With Zip Ties
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 2/19 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suture (N=19) | Adhesive Wound Closure Device (N=19) | Adhesive Wound Closure Device With Zip Ties (N=18)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT05251064/Prot_SAP_001.pdf
  • Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT05251064/ICF_000.pdf